CLINICAL TRIAL: NCT04456465
Title: Clinical Characteristics and Treatment of Pain Diabetic Peripheral Neuropathy（DPN） in China: a Multi-center Cross-sectional Survey
Brief Title: Pain Diabetic Peripheral Neuropathy（DPN) in China
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUTH2018054
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Diabetic Neuropathies
Keywords: Pain diabetic peripheral neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pain diabetic peripheral neuropathy — Neuropathic pain is the focus of current clinical research, clinical identification, and treatment. It is unique from nociceptive pain and requires evaluation of the relevance and utility of common pain measures created for other painful conditions.

SUMMARY:
To understand the clinical characteristics of DPN patients in China; To investigate the distribution of DPN patients with depression and anxiety symptoms; To investigate the related factors of moderate and severe pain in DPN patients; To investigate the treatment of pain and depression and/or anxiety in DPN patients.

DETAILED DESCRIPTION:
Pain diabetic peripheral neuropathy (DPN) is a heavy global economic burden. An American observational study in 2013 showed that the total average annual adjusted direct medical cost/person for DPN patients was $4,841, and the total average annual adjusted indirect medical cost/person was $9,730. A retrospective study in the United States in 2015 showed that the total annual direct medical cost per person for diabetes was $6,632, DPN ($12,492), DPN ($27,931), and severe DPN ($30,755) were 4.6 times higher than those for patients with diabetes alone. According to the 2015 European survey, the total annual direct medical cost per person for DPN patients in the United Kingdom was €2,963 (£2,511), of which 40% was used for hospitalization.

At present, there are no studies on the population epidemiology, depression and drug use of DPN in China. This study mainly investigates the above problems.

ELIGIBILITY:
Inclusion Criteria:

* outpatients who are elder than 18 years old with history of type 1or type 2 diabetes
* The presence of symptoms, signs and/or electrophysiological evidence of diabetic peripheral neuropathy
* The patient presents spontaneous pain (continuous or intermittent acupuncture pain, electric shock pain, burning pain, etc.) or induced pain (sensory hypersensitivity, paresthesia, etc.)
* The pain lasts for at least 3 months
* Informed consent has been signed

Exclusion Criteria:

* Patients with other causes of neuropathic, non-neuropathic, or mixed pain: for example, cervical/lumbar degenerative diseases, arthritis, nerve root compression, paraneoplastic syndromes, cerebrovascular diseases, spinal diseases, other peripheral neuropathies (immunological, toxic, nutritional peripheral neuropathies, etc.)
* Dementia, substance abuse, etc., severely affect cognitive and communication skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pain diabetic peripheral neuropathy（DPN） in China
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
moderate and severe pain (VAS score ≥4) | Time at recruitment
  The correlation factors of moderate and severe pain (VAS score ≥4) were analyzed exploratively. A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Demographic data | Time at recruitment
  A history of diabetes, diabetic peripheral neuropathy, and pain diabetic peripheral neuropathy Comorbidities such as hypertension, cardiovascular disease, a history of depressive disorders
Clinical manifestations of pain: VAS score | Time at recruitment
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. A higher score indicates greater pain intensity.
Depression screening/assessment: PHQ-9 scale | Time at recruitment
  The Patient Health Questionnaire (PHQ)-9 is the major depressive disorder (MDD) module of the full PHQ. Scores each of the criteria of MDD as "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score.
Anxiety screening/assessment: GAD-7 scale | Time at recruitment
  Generalized Anxiety Disorder 7-Item Scale (GAD-7): This symptom assessment tool measures seven anxiety symptoms on 4-point scales. Average time to complete: 3 minutes. Interpretation: Total scores of 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, MD.PHD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No